CLINICAL TRIAL: NCT04424758
Title: Testing Video Information About Mammography Screening in a Randomized Design
Brief Title: Testing Video Information About Mammography Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Manja Dahl Jensen, Principal investigator, Medical doctor, PhD-student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2204MDJ
Record Dates: First submitted 2020-05-28; First posted 2020-06-11 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: See protocol
Who Masked: Investigator, Outcomes Assessor
Masking Description: See protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receives information about mammography screening through a video. The video was developed with the goal of informing about mammography screening in a societal perspective using best available evidence.
  Interventions: Other: Video information about mammography screening
- Control group (Placebo Comparator): Receives information about energy systems through a video. The video does not contain any information related to mammography screening.
  Interventions: Other: Video information about smart energy systems

INTERVENTIONS:
Other: Video information about mammography screening — A video informing about mammography screening
  Arms: Intervention group
Other: Video information about smart energy systems — A video informing about smart energy systems
  Arms: Control group

SUMMARY:
This study examines how video information about mammography screening effect participants knowledge opinions and choice about screening.

DETAILED DESCRIPTION:
This study will be conducted as a single site parallel-arm, 1:1 randomized controlled trial (RCT) through a web-based quantitative survey uploaded in online forums. Participants will be randomized to either the intervention group (video information about mammography screening followed by a survey about mammography screening) or the control group (video information about energy systems followed by the same survey). The survey computer programme will randomly assign each respondent to either the intervention arm or the control arm in the beginning of the survey.

The allocation will be concealed from the researchers. The survey computer programme will deliver the intervention right after randomization. Participants will be aware of the allocation. However, they do not know about the study design. Data analysts will be kept blinded to the allocation.

Choice, knowledge and opinions related to mammography screening will be compared between the control group and the intervention group at one timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for the study includes all men and women age 18-75.

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Choice: proportion of participants in favor of mammography screening | One month
  The primary outcome in the study is choice. A possible effect of the intervention on choice will be examined by comparing the proportion of participants in favor of screening (on the individual level and societal level respectively) between the intervention arm and the control arm. One question addressing the societal choice and one question addressing the individual choice is included in our questionnaire.

SECONDARY OUTCOMES:
Response duration: time | One month
  Response duration is registered for all participants in the online survey. Mean response duration will be calculated in both the intervention arm and control arm.
Acceptability of the video: percentage of participants finding the video to be neutral, in favor of or against mammography screening. | One month
  Percentages of the participants finding the video to be neutral, in favor of or against mammography screening will be calculated in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Manja Jensen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Section of General Practice, Copenhagen, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed, access to study data will be provided by the PI on request.
Supporting Information: Study Protocol
Time Frame: Data will be stored until 2050.
Access Criteria: Data will be provided by the PI on request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04424758/Prot_SAP_000.pdf